CLINICAL TRIAL: NCT03728101
Title: A Clinical Trial to Evaluate the Effect of Simvastatin on the Pharmacokinetics and Pharmacodynamics of Dabigatran in Healthy Male Adults
Brief Title: Drug Interaction Study of Simvastatin and Dabigatran
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyewon Chung, Clinical instructor, Korea University Guro Hospital
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SD-DDI
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — Simvastatin; Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): * Dabigatran etexilate
  * Simvastatin + Dabigatran etexilate
  Interventions: Drug: Simvastatin, Dabigatran Etexilate

INTERVENTIONS:
Drug: Simvastatin, Dabigatran Etexilate — The subjects receive dabigatran etexilate with and without simvastatin administration

SUMMARY:
The aim of the study is to evaluate the effect of simvastatin on the pharmacokinetics and pharmacodynamics of dabigatran in healthy male adults

DETAILED DESCRIPTION:
Pharmacokinetics and pharmacodynamics of dabigatran without coadministration of simvastatin will be compared with those after multiple administration of simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 19 and 50 years
* Subjects with body mass index (BMI) between 18.5 and 29.9 kg/m2 and weight more than 50 kg
* Subjects who agree with performing contraception during the study
* Subjects who agreed with written informed consent

Exclusion Criteria

* Subjects who have a current or prior history of cardiovascular, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, skin, psychiatric, or neurological diseases that is clinically significant
* Subjects who have clinically significant allergic history or allergy to simvastatin, dabigatran, or other components of drug
* Creatinine clearance is below 60 ml/min
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) is more than 2-fold of upper limit or normal range
* Subjects who have clinically significant bleeding
* Subjects at risk of bleeding
* Subjects who took drugs which significantly interact with simvastatin or dabigatran prior to dosing
* Whole blood donation within 60 days prior to dosing, or apheresis donation within 20 days prior to dosing
* Participated in a previous clinical trial within 90 days prior to dosing
* Subjects with a history of alcohol abuse
* Subjects who are determined by investigator's decision as unsuitable for clinical trial participation

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Cmax | 24 hours
  maximum plasma concentration
AUC | 24 hours, zero to infinite
  Area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
aPTT | 24 hours
  Activated partial thromboplastin time
TT | 24 hours
  Thrombin time
lag time | 24 hours
  thrombin generation assay
peak thrombin | 24 hours
  thrombin generation assay
velocity index | 24 hours
  thrombin generation assay
area under the curve | 24 hours
  thrombin generation assay

CONTACTS AND LOCATIONS:
Overall Officials: Hyewon Chung, MD, PhD, Principal Investigator — Clinical Instructor
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea